CLINICAL TRIAL: NCT06395831
Title: Assessment of Quality of Life and Independence, as Well as Received Social Support in Patients Before and After Surgery for Spinal Cancer
Brief Title: Assessment of Quality of Life and Independence, as Well as Received Social Support for Spinal Cancer.
Status: Recruiting | Type: Observational
Sponsor: Andrzej Frycz Modrzewski Krakow University (Other)
Responsible Party: Principal Investigator, Edyta Laska, Principal Investigator, Andrzej Frycz Modrzewski Krakow University
Other Study IDs: 32/2023
Record Dates: First submitted 2024-01-01; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Spinal Canal Tumors
MeSH Terms: conditions — Spinal Cord Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: BREF,ADL,AIS — 1. abbreviated version of the quality of life assessment questionnaire - The World Health Organization Quality of Life (WHOQOL) -BREF
  2. scale I - ADL according to Lawton
  3. the AIS questionnaire
  4. the Zimet Multidimensional Scale of Perceived Social Support - the original version of the MSPSS

SUMMARY:
* Evaluation of the quality of life of patients before and after surgery for benign and malignant spinal cancers, assessing whether it depends on the size of the tumor, type of cancer, malignancy and its location
* evaluation of patients' independence before and after surgery for benign and malignant spinal tumors, evaluation of what factors influenced patients' different independence
* multidimensional assessment of perceived social support of patients before and after surgery for benign and malignant spinal cancers, taking into account three sources of support: significant person, family and friends

DETAILED DESCRIPTION:
RESEARCH PROJECT DESCRIPTION, RESEARCH METHODOLOGY:

Research objectives:

* To evaluate the quality of life of patients before and after surgery for benign and malignant spinal cancers, to assess whether it depends on the size of the tumor, type of cancer, malignancy and its location
* evaluation of patients' independence before and after surgery for benign and malignant spinal tumors, assessment of what factors influenced patients' different independence
* multidimensional evaluation of perceived social support of patients before and after surgery for benign and malignant spinal cancers, taking into account three sources of support: significant person, family and friends

Scientific (research) problems:

* What is the quality of life of patients before and after surgery for benign and malignant spinal cancers ? Is the quality of life in patients with spinal cancer dependent on tumor size, malignancy, location or type of cancer ?
* How do patients rate their independence both before and after surgery for spinal cancers at different stages of the disease?
* How do patients with spinal cancer at different stages of the disease rate the social support they received both before and after surgery?

ELIGIBILITY:
Inclusion criteria for the study:

-clinical diagnosis of spinal cancer

Study exclusion criteria:

-inflammatory and disc disease of the spinal column

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Each patient who is admitted to the surgical ward with a diagnosis of spinal cancer will be qualified for surgery will be given written consent for the study and the processing of personal data, as well as information for the researcher with questionnaires, and will then give written consent and be recruited for the study. The patient's personal data processing information will be retained for the study until its completion.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life assessed using The World Health Organization Quality of Life (WHOQOL) scale. Social support assessed using Zimet's Multidimensional Perceived Social Support Scale - the original version on the MSPSS. | 12 months to 24 months
  Quality of life assessed using The World Health Organization Quality of Life (WHOQOL-BREF) scale questionnaire which contains 26 questions analyzing four domains of life and separately perception of quality of life and self-assessment of health status.
  It is used to assess the quality of life of both healthy and sick people in clinical practice and addresses the following domains of quality of life: somatic functioning, psychological functioning, social functioning and community functioning.
  Social support assessed using Zimet's Multidimensional Perceived Social Support Scale - the original version on the MSPSS.
  The Multidimensional Scale of Perceived Social Support takes into account the multidimensionality of perceived social support, considering three primary sources of support: significant other, family and friends. The scale consists of 12 statements, which the subject addresses using a seven-point Likert scale, where 1 means "strongly disagree" and 7 means "strongly agree."

CONTACTS AND LOCATIONS:
Locations (1):
- St. Raphael's Hospital, Krakow, Lesserpoland, Poland

IPD SHARING:
Plan to Share IPD: No